CLINICAL TRIAL: NCT03007147
Title: International Phase 3 Trial in Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia (Ph+ALL) Testing Imatinib in Combination With Two Different Cytotoxic Chemotherapy Backbones
Brief Title: Imatinib Mesylate and Combination Chemotherapy in Treating Patients With Newly Diagnosed Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: EsPhALL (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL1631; NCI-2016-01588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL1631; 2017-000705-20; AALL1631 (Other: Children's Oncology Group); AALL1631 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia; Mixed Phenotype Acute Leukemia; T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Stem Cell Transplantation; calaspargase pegol; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Dexrazoxane; Razoxane; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Ifosfamide; Imatinib Mesylate; Leucovorin; Levoleucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; Methylprednisolone; exifone; Medrol Veriderm; pegaspargase; Prednisolone; Hydrocortisone; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (imatinib mesylate, EsPhALL chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Dexrazoxane Hydrochloride; Drug: Doxorubicin; Drug: Etoposide; Biological: Filgrastim; Drug: Ifosfamide; Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Levoleucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Drug: Prednisolone; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm B (imatinib mesylate, COG/BFM chemotherapy) (Experimental): See Detailed Description.
  Interventions: Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Dexrazoxane Hydrochloride; Drug: Doxorubicin; Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Levoleucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Drug: Prednisolone; Other: Questionnaire Administration; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT) (Experimental): See Detailed Description
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Dexrazoxane Hydrochloride; Drug: Doxorubicin; Drug: Etoposide; Biological: Filgrastim; Drug: Ifosfamide; Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Levoleucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Drug: Prednisolone; Other: Questionnaire Administration; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
  Arms: Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT)
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IV, SC, or IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: Arm A (imatinib mesylate, EsPhALL chemotherapy); Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Dexrazoxane Hydrochloride — Given IV
  Other Names: Cardioxane; Totect; Zinecard
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: Arm A (imatinib mesylate, EsPhALL chemotherapy); Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT)
Biological: Filgrastim — Given SC or IV
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
  Arms: Arm A (imatinib mesylate, EsPhALL chemotherapy); Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT)
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Arm A (imatinib mesylate, EsPhALL chemotherapy); Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT)
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP 57148B; CGP-57148; CGP-57148B; CGP57148; CGP57148B; Gleevec; Glivec; Imarech; Imat; Imkeldi; STI 571; STI-571; STI571
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given PO or IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Levoleucovorin — Given PO or IV
  Other Names: CL-307,782; Elvorine, Isovorin, Levofolene, Levorin; Isovorin; L-Leucovorin; Levofolinate; Levofolinic acid
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Arm A (imatinib mesylate, EsPhALL chemotherapy); Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT)
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisolone — Given PO
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
Other: Questionnaire Administration — Ancillary studies
Drug: Therapeutic Hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid
  Arms: Arm A (imatinib mesylate, EsPhALL chemotherapy); Arm C (imatinib mesylate, EsPhALL chemotherapy, HSCT)
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase III trial studies how well imatinib mesylate works in combination with two different chemotherapy regimens in treating patients with newly diagnosed Philadelphia chromosome positive acute lymphoblastic leukemia (ALL). Imatinib mesylate has been shown to improve outcomes in children and adolescents with Philadelphia chromosome positive (Ph+) ALL when given with strong chemotherapy, but the combination has many side effects. This trial is testing whether a different chemotherapy regimen may work as well as the stronger one but have fewer side effects when given with imatinib. The trial is also testing how well the combination of chemotherapy and imatinib works in another group of patients with a type of ALL that is similar to Ph+ ALL. This type of ALL is called "ABL-class fusion positive ALL", and because it is similar to Ph+ ALL, is thought it will respond well to the combination of agents used to treat Ph+ ALL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare disease-free survival (DFS) of standard risk (SR) pediatric Philadelphia chromosome (Ph)+ acute lymphoblastic leukemia (ALL) treated with continuous imatinib mesylate (imatinib) combined with either a high-risk Children's Oncology Group (COG) ALL chemotherapy backbone or the more intensive European (Es)PhALL chemotherapy backbone.

SECONDARY OBJECTIVES:

I. To compare DFS of SR pediatric Ph+ and ABL-class fusion positive ALL patients treated with continuous imatinib combined with either a high-risk COG-ALL chemotherapy backbone or the more intensive EsPhALL chemotherapy backbone.

II. To determine the feasibility of administration of imatinib after allogeneic hematopoietic stem cell transplantation (HSCT) in high risk (HR) Ph+ ALL patients.

III. To determine event-free survival (EFS) of HR pediatric Ph+ ALL patients treated with EsPhALL chemotherapy, HSCT in first complete remission and post-HSCT imatinib.

IV. To compare rates of grade 3 or higher infections in standard risk (SR) Ph+ ALL patients between the two randomized arms.

V. To evaluate EFS and overall survival (OS) of all eligible Ph+ALL patients enrolled on the study.

VI. To evaluate OS in SR Ph+ ALL patients. VII. To evaluate OS in HR Ph+ ALL patients. VIII. To evaluate EFS and OS of all eligible ABL-class fusion positive ALL patients enrolled on the study.

EXPLORATORY OBJECTIVES:

I. To describe the toxicities associated with post-HSCT administration of imatinib in HR Ph+ALL patients.

II. To evaluate the long-term toxicities in SR Ph+ ALL patients treated with chemotherapy plus imatinib (no transplant), overall and between both randomized arms.

III. To determine prognostic significance of minimal residual disease (MRD) in Ph+ ALL at various time points during therapy.

IIIa. To evaluate MRD in HR patients just prior to HSCT and then at regular intervals post-HSCT and explore the association of these measurements with long-term outcome.

IIIb. To evaluate concordance of MRD assessments made by IGH-T cell receptor (TCR) polymerase chain reaction (PCR) assay and next generation sequencing (NGS) assays.

IV. To determine and validate if IKZF1 deletions alone (IKZF1del) or with other transcription factor deletions (ie, IKZF1 plus subtype [IKZF1plus]) or other identified genetic lesions predict poor outcomes in Ph+/ABL-class Ph-like ALL in patients treated on AALL1631.

V. To determine the frequency and prognostic significance of p190 and p210 BCR::ABL1 fusion variants in pediatric Ph+ ALL/ABL-class Ph-like ALL.

VI. To measure adherence to oral chemotherapeutic agents (imatinib, 6-mercaptopurine and methotrexate) during the maintenance phase in SR Ph+ ALL patients.

VIa. To identify factors associated with poor adherence. VIb. To determine association between relapse risk and adherence to each oral chemotherapeutic agent (separately and combined).

VII. To measure adherence to imatinib after allogeneic HSCT in HR Ph+ ALL patients and identify factors associated with poor adherence.

VIII. To compare DFS of SR ABL-class fusion positive ALL patients treated with continuous imatinib combined with either a high-risk COG-ALL chemotherapy backbone or the more intensive EsPhALL chemotherapy backbone.

IX. To determine the potential therapeutic impact of major secondary events via pharmacologic inhibitor screens in existing/engineered cell models of Ph+ and ABL-class Ph-like ALL harboring secondary events and to test the in vivo activity of the most compelling candidate compounds from pilot studies using patient-derived xenograft (PDX) models established from Ph+ and ABL-class Ph-like ALL samples collected from patients treated on AALL1631.

X. To decipher the molecular and cellular heterogeneity of chronic myelogenous leukemia (CML)-like versus typical Ph+ ALL via single-cell genomics and functional assays and investigate CML-like phenotypes via single-cell ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) sequencing to identify distinct transcriptomic and mutational profiles that will provide novel opportunities for diagnostic and therapeutic interventions.

OUTLINE:

INDUCTION IA PART 1: Patients receive induction IA according to standard of care on days 1-14.

INDUCTION IA PART 2: Patients receive imatinib mesylate orally (PO) once daily (QD) or twice daily (BID) on days 15-33, prednisolone PO twice daily (BID) or methylprednisolone intravenously (IV) on days 15-28, vincristine sulfate IV over 1 minute on days 15 and 22, daunorubicin hydrochloride IV over 1-15 minutes on days 15 and 22, and methotrexate intrathecally (IT) on day 29.

INDUCTION IB: Patients receive imatinib mesylate PO QD or BID on days 1-35, cyclophosphamide IV over 30-60 minutes on days 1 and 28, mercaptopurine PO on days 1-28, cytarabine IV or subcutaneously (SC) on days 3-6, 10-13, 17-20, and 24-27, and methotrexate IT on days 10 and 24.

POST-INDUCTION THERAPY: Patients classified as standard risk are randomized to 1 of 2 arms. Patients with high risk are assigned to Arm C.

ARM A:

CONSOLIDATION BLOCK 1: Patients receive imatinib mesylate PO QD or BID on days 1-21, methotrexate IT, cytarabine IT, and therapeutic hydrocortisone IT on day 1, high dose methotrexate IV over 24 hours on day 1, vincristine sulfate IV over 1 minute on days 1 and 6, dexamethasone PO BID or IV on days 1-5, cyclophosphamide IV over 30-60 minutes on days 2-4, leucovorin calcium or levoleucovorin PO or IV on days 3 and 4, high dose cytarabine IV over 3 hours and pegaspargase or calaspargase pegol IV over 1-2 hours on day 5, and filgrastim SC or IV on days 7-11 in the absence of disease progression or unexpected toxicity.

CONSOLIDATION BLOCK 2: Patients receive imatinib mesylate PO QD or BID on days 1-21, methotrexate IT, cytarabine IT, and therapeutic hydrocortisone IT on day 1, high dose methotrexate IV over 24 hours on day 1, dexamethasone PO BID or IV on days 1-5, vincristine sulfate IV over 1 minute on days 1 and 6, ifosfamide IV over 1 hour on days 2-4, leucovorin calcium or levoleucovorin PO or IV on days 3 and 4, dexrazoxane hydrochloride IV over 15 minutes and daunorubicin hydrochloride IV over 1-15 minutes on day 5, pegaspargase or calaspargase pegol IV over 1-2 hours on day 6, and filgrastim SC or IV on days 7-11 in the absence of disease progression or unexpected toxicity.

CONSOLIDATION BLOCK 3: Patients receive imatinib mesylate PO QD or BID on days 1-21, high dose cytarabine IV over 3 hours on days 1-3, dexamethasone PO BID or IV on days 1-5, etoposide IV over 1-2 hours on days 3-5, methotrexate IT, cytarabine IT, and therapeutic hydrocortisone IT on day 5, pegaspargase or calaspargase pegol IV over 1-2 hours on day 6, and filgrastim SC or IV on days 7-11 in the absence of disease progression or unexpected toxicity.

DELAYED INTENSIFICATION 1 PART 1: Patients receive imatinib mesylate PO QD or BID on days 1-35, methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine sulfate IV over 1 minute, dexrazoxane hydrochloride IV over 15 minutes, and doxorubicin IV over 3-15 minutes on days 8, 15, 22, and 29, and pegaspargase or calaspargase pegol IV over 1-2 hours on day 8 in the absence of disease progression or unexpected toxicity.

DELAYED INTENSIFICATION 1 PART 2: Patients receive imatinib mesylate PO QD on days 36-63, cyclophosphamide IV over 30-60 minutes on day 36, thioguanine PO on days 36-49, cytarabine IV over 1-30 minutes or SC on days 38-41 and 45-48, and methotrexate IT on days 38 and 45in the absence of disease progression or unexpected toxicity.

INTERIM MAINTENANCE: Patients receive imatinib mesylate PO QD or BID on days 1-28, methotrexate PO on days 1, 8, 15, and 22, and mercaptopurine PO on days 1-28 in the absence of disease progression or unexpected toxicity.

DELAYED INTENSIFICATION 2 PART 1: Patients receive imatinib mesylate PO QD or BID on days 1-35, methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine sulfate IV over 1 minute, dexrazoxane hydrochloride IV over 15 minutes, and doxorubicin IV over 3-15 minutes on days 8, 15, 22, and 29, and pegaspargase or calaspargase pegol IV over 1-2 hours on day 8 in the absence of disease progression or unexpected toxicity.

DELAYED INTENSIFICATION 2 PART 2: Patients receive imatinib mesylate PO QD on days 36-49, cyclophosphamide IV over 30-60 minutes on day 36, thioguanine PO on days 36-49, cytarabine IV over 1-30 minutes or SC on days 36-39 and 43-46, and methotrexate IT on days 36 and 43 in the absence of disease progression or unexpected toxicity.

MAINTENANCE: Patients receive imatinib mesylate PO QD or BID on days 1-84, methotrexate PO once weekly (QW) and IT on days 1 and 43 of cycles 1, 2, and 3, and mercaptopurine PO on days 1-84. Cycles with imatinib mesylate and mercaptopurine repeat every 84 days for up to 104 weeks from the start of Induction IA in the absence of disease progression or unexpected toxicity.

ARM B:

INTERIM MAINTENANCE: Patients receive imatinib mesylate PO QD or BID on days 1-63, vincristine sulfate IV over 1 minute and high dose methotrexate IV over 24 hours on days 1, 15, 29, and 43, leucovorin calcium or levoleucovorin PO or IV on days 3-4, 17-18, 31-32, and 45-46, mercaptopurine PO on days 1-56, and methotrexate IT on days 1 and 29 in the absence of disease progression or unexpected toxicity.

DELAYED INTENSIFICATION PART 1: Patients receive imatinib mesylate PO QD or BID on days 1-28, methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine sulfate IV over 1 minute, dexrazoxane hydrochloride IV over 15 minutes, and doxorubicin IV over 3-15 minutes on days 1, 8, and 15, and pegaspargase or calaspargase pegol IV over 1-2 hours or IM on day 4 in the absence of disease progression or unexpected toxicity.

DELAYED INTENSIFICATION PART 2: Patients receive imatinib mesylate PO QD on days 29-56, cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39, methotrexate IT on days 29 and 36, vincristine sulfate IV over 1 minute on days 43 and 50, and pegaspargase or calaspargase pegol IV over 1-2 hours on day 43 in the absence of disease progression or unexpected toxicity.

INTERIM MAINTENANCE WITH CAPIZZI METHOTREXATE: Patients receive imatinib mesylate PO QD or BID on days 1-56, vincristine sulfate IV over 1 minute and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and pegaspargase or calaspargase pegol IV over 1-2 hours on days 2 and 23 in the absence of disease progression or unexpected toxicity.

MAINTENANCE: Patients receive imatinib mesylate PO QD or BID on days 1-84, vincristine sulfate IV over 1 minute on days 1, 29, and 57, prednisolone PO BID (or methylprednisolone IV for cycle 1 and 2) on days 1-5, 29-33, and 57-61, mercaptopurine PO on days 1-84, methotrexate PO QW, and methotrexate IT on day 1 (and day 29 for cycle 1 and 2). Cycles repeat every 84 days for up to 104 weeks from the start of Induction IA in the absence of disease progression or unexpected toxicity.

ARM C:

CONSOLIDATION BLOCK 1: Patients receive imatinib mesylate, methotrexate, cytarabine, therapeutic hydrocortisone, high dose methotrexate, vincristine sulfate, dexamethasone, leucovorin calcium or levoleucovorin, high dose cytarabine, and pegaspargase or calaspargase pegol as in Arm A Consolidation Block 1, and filgrastim SC or IV on day 7 in the absence of disease progression or unexpected toxicity.

CONSOLIDATION BLOCK 2: Patients receive imatinib mesylate, methotrexate, cytarabine, therapeutic hydrocortisone, high dose methotrexate, dexamethasone, vincristine sulfate, ifosfamide, leucovorin calcium or levoleucovorin, dexrazoxane hydrochloride, daunorubicin hydrochloride, pegaspargase or calaspargase pegol, and filgrastim as Arm A Consolidation Block 2 in the absence of disease progression or unexpected toxicity.

CONSOLIDATION BLOCK 3: Patients receive imatinib mesylate, dexamethasone, etoposide, methotrexate, cytarabine, therapeutic hydrocortisone, pegaspargase or calaspargase pegol, and filgrastim as in Arm A Consolidation Block 3, and high dose cytarabine IV over 3 hours on days 1-2 in the absence of disease progression or unexpected toxicity.

HSCT: Patients undergo HSCT on day 0. Patients who do not proceed to HSCT receive Delayed Intensification 1, Interim Maintenance, Delayed Intensification 2, and Maintenance as in Arm A.

POST-HSCT: Patients receive imatinib mesylate PO QD or BID starting on days 56-365 in the in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up every year for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* For patients enrolled on APEC14B1 prior to enrollment on AALL1631, the required diagnostic bone marrow sample has been fulfilled

  * For patients who have not previously enrolled on APEC14B1 prior to enrollment on AALL1631, a baseline diagnostic sample (or peripheral blood sample with blasts if marrow sample unavailable) must be available to develop an MRD probe
  * In addition, laboratory reports detailing evidence of BCR::ABL1 fusion or ABL-class fusion must be submitted for rapid central review within 72 hours of study enrollment
* >= 1 year (365 days) and =< 21 years at ALL diagnosis
* Ph+ (BCR::ABL1 fusion): newly diagnosed de novo ALL (B-ALL or T-ALL) or mixed phenotypic acute leukemia (MPAL meeting 2016 World Health Organization [WHO] definition) with definitive evidence of BCR::ABL1 fusion by karyotype, fluorescence in situ hybridization (FISH) and/or molecular methodologies
* ABL-class fusion: newly diagnosed B-ALL with definitive evidence of ABL-class fusions. ABL-class fusions are defined as those involving the following genes: ABL1, ABL2, CSF1R, PDGFRB, PDGFRA. Methods of detection include fluorescence in-situ hybridization ([FISH], e.g. using break-apart or colocalization signals probes), multiplex or singleplex reverse-transcription polymerase chain reaction (RT-PCR), whole transcriptome or panel-based RNA-sequencing (e.g. TruSight RNA Pan-Cancer Panel; Illumina, San Diego, California [CA], United States of America [USA] or similar)
* Ph+ patients must have previously started Induction therapy, which includes vincristine, a corticosteroid, pegaspargase, with or without anthracycline, and/or other standard cytotoxic chemotherapy
* Ph+ patients have not received more than 14 days of multiagent Induction therapy beginning with the first dose of vinCRIStine
* Ph+ patients may have started imatinib prior to study entry but have not received more than 14 days of imatinib
* ABL-class fusion patients must have previously completed the 4 or 5 weeks of multiagent Induction chemotherapy (Induction IA phase)
* ABL-class fusion patients may have started imatinib during Induction IA, at the same time of or after the first vinCRIStine dose
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2
* Direct bilirubin =< 2.0 mg/dL
* Shortening fraction of >= 27% by echocardiogram
* Ejection fraction of >= 50% by radionuclide angiogram or echocardiogram
* Corrected QT interval, QTc < 480 msec

  * Note: Repeat echocardiogram and electrocardiogram are not required if they were performed at or after initial ALL diagnosis, before study enrollment
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or serum creatinine within normal limits based on age/gender, as follows:

  * 1 to < 2 years: maximum serum creatinine 0.6 mg/dL (both male and female)
  * 2 to < 6 years: maximum serum creatinine 0.8 mg/dL (both male and female)
  * 6 to < 10 years: maximum serum creatinine 1 mg/dL (both male and female)
  * 10 to < 13 years: maximum serum creatinine 1.2 mg/dL (both male and female)
  * 13 to < 16 years: maximum serum creatinine 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: maximum serum creatinine 1.7 mg/dL (male), 1.4 mg/dL (female)

Exclusion Criteria:

* Known history of chronic myelogenous leukemia (CML)
* ALL developing after a previous cancer treated with cytotoxic chemotherapy
* Active, uncontrolled infection, or active systemic illness that requires ongoing vasopressor support or mechanical ventilation
* Down syndrome
* Pregnancy and breast feeding

  * Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
  * Lactating females who plan to breastfeed their infants
  * Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of treatment according to protocol
* Patients with congenital long QT syndrome, history of ventricular arrhythmias or heart block
* Prior treatment with dasatinib, or any TKI other than imatinib

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 475 (Estimated)
Dates: Start 2017-08-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) of Randomized Arms (standard risk [SR] Philadelphia chromosome [Ph+] acute lymphoblastic leukemia [ALL] patients) | Up to 3 years
  Three-year DFS and 95% confidence intervals (CI) of SR Ph+ ALL patients treated continuous imatinib mesylate with high risk Children's Oncology Group (COG)-ALL chemotherapy backbone or more intensive European (Es)PhALL chemotherapy backbone.

SECONDARY OUTCOMES:
DFS on Randomized Arms (SR Ph+ ALL and ABL-class fusion positive patients) | Up to 3 years
  Three-year DFS (time from randomization to relapse, second malignancy, or death in complete remission) and 95% CI of SR pediatric Ph+ and ABL-class fusion positive patients treated with continuous imatinib combined with either a high-risk COG-ALL chemotherapy backbone or the more intensive EsPhALL chemotherapy backbone.
Feasibility of post hematopoietic stem cell transplantation (HSCT) imatinib mesylate administration after allogenic HSCT in high risk Ph+ ALL patients | Up to 2 years
  The proportion of patients who receive at least 75% of intended doses.
Event free survival (EFS) of high risk pediatric Ph+ ALL patients treated with EsPhALL chemotherapy, HSCT in first complete remission, and post-HSCT imatinib mesylate | Up to 3 years
  Three-year EFS and 95% CI for high risk pediatric Ph+ ALL patients treated with EsPhALL chemotherapy, HSCT in first complete remission, and post-HSCT imatinib mesylate. EFS is defined as the time from the date of bone marrow for minimal residual disease (MRD) assessment at end-IB to first event (resistant disease [MRD >= 10-2 or morphologic residual disease at end of consolidation block 3], relapse, progressive disease [i.e., MRD >= 10-2 at two post-HSCT time points separated by at least 2 weeks], second malignancy, or death in complete remission), or time to last follow-up for patients without events.
Incidence of grade 3 or higher infections in standard risk Ph+ ALL patients in the two randomized arms | Up to 3 years
  Evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The rate of infections during the post IB/pre-maintenance phases of treatment will be described for each randomization group.
EFS of all Ph+ patients | Up to 3 years
  Three-year EFS and 95% CI for Ph+ ALL patients. EFS here is defined as the time from enrollment until resistant disease, relapse, progressive disease post-HSCT, second malignant, or death, whichever occurs first.
Overall survival (OS) of all Ph+ patients | Up to 3 years
  Three-year OS and 95% CI for Ph+ ALL patients. OS is defined as the time from study enrollment to death from any cause.
OS of SR Ph+ patients | Up to 3 years
  Three-year OS (time from randomization to death from any cause) and 95% CI of SR pediatric Ph+ patients
OS of SR Ph+ patients by randomization group | Up to 3 years
  Three-year OS (time from randomization to death from any cause) and 95% CI of SR pediatric Ph+ patients by randomization group: treated with continuous imatinib combined with either a high-risk COG-ALL chemotherapy backbone or the more intensive EsPhALL chemotherapy backbone.
OS of high risk Ph+ patients | Up to 3 years
  Three-year OS (time from the date of MRD assessment at end-IB to death from any cause) and 95% CI of HR pediatric Ph+ patients.
EFS of all eligibility ABL-class fusion positive ALL patients | Up to 3 years
  Three-year EFS (time from enrollment until resistant disease, relapse, progressive disease post-HSCT, second malignancy, or death, whichever occurs first) and 95% CI of ABL-class fusion positive patients.
OS of all eligibility ABL-class fusion positive ALL patients | Up to 3 years
  Three-year OS (the time from study enrollment to death from any cause) and 95% CI of ABL-class fusion positive patients.

OTHER OUTCOMES:
Incidence of toxicities associated with post-HSCT administration of imatinib mesylate | Up to 2 years
  Evaluated according to NCI CTCAE version 5.0. Frequencies of target toxicities in high risk patients after the initiation of post-HSCT imatinib mesylate will be described. For the high risk patients, the specific targeted toxicities will include grade 4 neutropenia, grade 4 thrombocytopenia, grade 3 or higher bilirubin, grade 4 or higher transaminitis, and grade 3 or higher infection.
Incidence of long-term toxicities in patients treated with chemotherapy plus imatinib mesylate (no transplant) in both arms | Up to 3 years
  Evaluated according to NCI CTCAE version 5.0. Frequencies of long-term toxicities will be described and differences between randomized arms will be explored. Specific long-term toxicities to be explored include cardiac (echocardiographic abnormalities, including decreased left ventricular (LV) function and decreased LV wall thickness), growth (linear height, bone age), and second malignant neoplasm.
MRD measured by IGH-T cell receptor (TCR) polymerase chain reaction (PCR) and next generation sequencing (NGS) assay | Up to 6 months
  For all patients, frequencies and prognostic significance (DFS, EFS, OS) will be explored for MRD levels (i.e., MRD negative, detectable at < 5 x 10^-4, and dectectable at >= 5 x 10^-4) at end of Induction IB.
MRD in high risk Ph+ patients measured by IGH-TCR PCR and NGS assay | Up to 3 years
  The outcome of high risk Ph+ patients will be described, including proportion of patients who achieve MRD-negativity just prior to HSCT, and at regular intervals post-HSCT. Associations between these findings and long-term outcomes (e.g., OS, DFS) will be explored.
MRD assessments made by IGH-TCR PCR assay and NGS assay | Up to 3 years
  Concordance of MRD assessments made by IGH-TCR PCR assay and NGS assay will be described and evaluated. Scatter plots and diagrams will be used to examine agreements and patterns of agreement or any differences found. Concordance will be explored both for the overall cohort, as well as by risk group. The increased sensitivity of the NGS will be closely examined to find cases where the MRD levels are detectable by NGS but undetectable by PCR, as well as cases in which one test yields results and the other does not (test failure). Prognostic relationships on outcomes for these subjects will be inspected.
IKZF1 deletions alone | Up to 3 years
  Will determine and validate if IKZF1 deletions alone predict poor outcomes in Ph+/ABL-class Ph-like ALL in patients treated on AALL1631.
IKZF1 deletions with other transcription factor deletions | Up to 3 years
  Will determine and validate if IKZF1 deletions with other transcription factor deletions predict poor outcomes in Ph+/ABL-class Ph-like ALL in patients treated on AALL1631.
Other identified genetic lesions | Up to 3 years
  Will determine and validate if other identified genetic lesions predict poor outcomes in Ph+/ABL-class Ph-like ALL in patients treated on AALL1631.
Frequency of p190 and p210 BCR::ABL1 fusion variants | Up to 3 years
  For both standard risk and high risk groups, frequencies and prognostic significance (OS, DFS) will be explored for p190 and p210 BCR::ABL1 fusion variants in pediatric Ph+ ALL/ABL-class Ph-like ALL.
Adherence to oral chemotherapeutic agents in standard risk Ph+ ALL patients | Up to 2 years
  Adherence to imatinib mesylate, 6-mercaptopurine, and methotrexate will be evaluated in COG-enrolled participants using an electronic monitoring device. Adherence rate will be computed for each month of adherence monitoring. Longitudinal binomial regression will be conducted using generalized estimating equation methods by modeling monthly adherence rate as an unstructured mean model using five indicator variables of time for the study months. Time in months will also be treated as a continuous variable to explore temporal trends in adherence rate. Compound symmetry will be assumed as the working correlation matrix over time. Covariates that will be considered for adjustment include those hypothesized to be predictors of adherence, annual household income, parental education, time since start of maintenance, risk classification for ALL, and imatinib, 6-mercaptopurine (6MP), and methotrexate dose-intensity.
Adherence to imatinib mesylate after allogeneic HSCT in high risk Ph+ ALL patients | Up to 2 years
  Longitudinal binomial regression will be conducted using generalized estimating equation methods by modeling monthly adherence rate as an unstructured mean model using five indicator variables of time for the study months. Time in months will also be treated as a continuous variable to explore temporal trends in adherence rate. Compound symmetry will be assumed as the working correlation matrix over time. Covariates that will be considered for adjustment include those hypothesized to be predictors of adherence, annual household income, parental education, time since start of maintenance, risk classification for ALL, and imatinib, 6MP, and methotrexate dose-intensity.
Therapeutic impact of major secondary events | Up to 3 years
  Will determine the potential therapeutic impact of major secondary events via pharmacologic inhibitor screens in existing/engineered cell models of Ph+ and ABL-class Ph-like ALL harboring secondary events.
In vivo activity | Up to 3 years
  Will test the in vivo activity of the most compelling candidate compounds from pilot studies using patient-derived xenograft models established from Ph+ and ABL-class Ph-like ALL samples collected from patients treated on AALL1631.
Molecular heterogeneity | Up to 3 years
  Will decipher the molecular heterogeneity of chronic myelogenous leukemia (CML)-like versus typical Ph+ ALL via single-cell genomics and functional assays.
Cellular heterogeneity | Up to 3 years
  Will decipher the cellular heterogeneity of CML-like versus typical Ph+ ALL via single-cell genomics and functional assays.
CML-like phenotypes | Up to 3 years
  Will investigate CML-like phenotypes via single-cell ribonucleic acid and deoxyribonucleic acid sequencing to identify distinct transcriptomic and mutational profiles that will provide novel opportunities for diagnostic and therapeutic interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Lewis B Silverman, Principal Investigator — Children's Oncology Group; Prof. Andrea Biondi, Principal Investigator — EsPhALL Network/ BFM Study Group
Locations (226):
- United States (184):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- St. Anna Children's Hospital, Vienna, Austria
- Hospitals Leuven, Leuven, Flemish Brabant, Belgium
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Hospital Roberto del Rio-Universidad de Chile, Santiago, Chile
- University Hospital Motol, Prague, Czechia
- Tampere University Hospital, Tampere, Finland
- CHU Hopital Sud, Rennes, France
- Germany (2):
  - University Medical Center chleswig- Campus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinik Eppendorf, Hamburg
- Hong Kong Children's Hospital, Kowloon Bay, Kowloon, Hong Kong
- Schneider Children's Medical Center of Israel, Petah Tikva, Central District, Israel
- Clinica Pediatrica Università Milano-Bicocca Ospedale S. Gerardo/Fondazione MBBM, Monza, Italy
- Princess Máxima Center for Pediatric Oncology, Utrecht, Netherlands
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (3):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- Skane University Hospital, Lund, Skåne County, Sweden
- University Children's Hospital, Zurich, Switzerland